CLINICAL TRIAL: NCT06072651
Title: Fundamental Biobehavioral Mechanisms Underlying the Integrated Development of Emotion, Attachment, and Nutritive Intake in the Mother-Infant Dyad
Brief Title: Mother-Baby Study - Relative Reinforcing Value (RRV)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Julie Lumeng, Thomas P Borders Family Research Professor of Child Behavior and Development, Professor of Pediatrics, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00227836 CT2; R01DK134979 (NIH)
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Eating Behavior
Keywords: eating behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Relative Reinforcing Value (Experimental): The researchers will enroll 150 children from the long-term observational study, NCT06039878.
  Interventions: Behavioral: Relative Reinforcing Value of Food

INTERVENTIONS:
Behavioral: Relative Reinforcing Value of Food — Researcher gives child opportunity to press a button to earn three types of rewards: a high-reward food, a low-reward food, and a non-food reward.

SUMMARY:
The study will test a model of biobehavioral mechanisms involved in the development of a system of emotion, attachment, and nutritive intake in the mother-infant dyad and the association of this system with maternal feeding behavior, child eating behavior, dietary intake, and adiposity.

To participate in this study the infant must also be enrolled in long-term observational study, NCT06039878.

DETAILED DESCRIPTION:
This interventional task is done with children while they are in the long-term observational study, NCT06039878, at approximately ages 18 and 36 months. In the observational study there are 300 participants (150 mothers and 150 children). In this trial only data from the children is collected and therefore only 150 participants are listed.

ELIGIBILITY:
The child is a participant in the observational study (NCT06039878).

Min Age: 0 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Relative Reinforcing Value (RRV) of food | Up to approximately 36 months
  The RRV is measured using the number of button presses for each reward type relative to other reward types

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lumeng, MD, Study Chair — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No